CLINICAL TRIAL: NCT06673849
Title: Effects of Rhythmic Stabilization Versus Ball Balancing on Upper Extremity Function in Children With Spastic Cerebral Palsy
Brief Title: Rhythmic Stabilization Versus Ball Balancing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/MASIFAH
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Spastic Cerebral Palsy (sCP)
Keywords: Ball Balancing; Corticobulbar tracts; Corticospinal tracts; Epilepsy; Rhythmic Stabilization; Spastic CP
MeSH Terms: conditions — Cerebral Palsy; Epilepsy

STUDY DESIGN:
Intervention Model Description: The study design will be a Randomized Clinical Trial in which non probability convenient sampling will be used. Two groups of 6-12 age will be formed in which participants will be randomly divided. Group A will receive Rhythmic Stabilization exercises and Group B will receive Ball Balancing.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic Stabilization group (Experimental): The CP child will positions his/her upper extremity anywhere in its available range of motion and holds an isometric contraction. The physiotherapist will provide enough resistance to cause the child to react, but not enough to break the isometric contraction. As the child progresses, length of time of rhythmic stabilization increases, the therapist's resistance increases, and amount of contact area between therapist's hands and child's upper extremity decreases. The exercise program consisted of 30-minute sessions per week for six weeks
  Interventions: Other: Rhythmic Stabilization
- Ball Balancing group (Experimental): Have the child balance on his/her hands on a 48-inch Gymnastic ball, first with eyes open, then closed. Progress from both hands on one large ball to each hand on separate balls and then to the weaker arm on one ball. Also, progress through the four body positions. With his/her eyes open, then closed. If he/she misses the position, he/she opens his/her eyes and actively moves to the desired position. Use a spotter, especially when doing this exercise for the first time or changing body positions, since the patient may fall off the Gymnastic ball. Start with one repetition of 10 seconds and progress to three to five repetitions of 60 seconds each and this will be done till 6 weeks
  Interventions: Other: Ball Balancing

INTERVENTIONS:
Other: Rhythmic Stabilization — Rhythmic Stabilization Program for Children with Cerebral Palsy Objective: Enhance upper extremity strength and stability through rhythmic stabilization exercises.
  Program Overview:
  Duration: 30-minute sessions Frequency: Once per week for 6 weeks
  Exercise Steps:
  Positioning: The child positions their upper extremity within their available range of motion.
  Isometric Contraction: The child holds an isometric contraction, maintaining the position without movement.
  Therapist's Role: Apply resistance that is sufficient to elicit a reaction but not enough to disrupt the isometric contraction.
  Progression: Gradually increase the duration of the isometric hold. Increase the amount of resistance applied. Decrease the contact area between the therapist's hands and the child's upper extremity to enhance stability challenges. Monitoring and Adjustments: Assess the child's ability to maintain the contraction and adapt the resistance and support as needed. Encourage the child's engagement.
  Arms: Rhythmic Stabilization group
Other: Ball Balancing — Ball Balancing Program Objective: Improve balance and stability. Equipment: 48-inch gymnastic ball
  Program Details:
  * Duration: 6 weeks
  * Frequency: As needed
  Steps:
  1. Initial Balance:
     * Eyes Open: Balance on hands for 10 seconds.
     * Progression: Increase to 3-5 repetitions of 60 seconds.
  2. Eyes Closed: Repeat the above exercise with eyes closed.
  3. Variations:
     * Both Hands on One Ball
     * Each Hand on Separate Balls
     * Weaker Arm on One Ball
  4. Body Positions: Progress through four body positions with eyes open, then closed.
  5. Correction: If the child misses a position, they open their eyes and reposition actively.
  Arms: Ball Balancing group

SUMMARY:
Spastic Cerebral Palsy (CP) is the leading cause of upper motor neuron syndrome (UMN) in children. The primary factors contributing to motor behavior disorders in these children are impairments in motor control and muscle strength. These impairments result in changes in muscle growth and hinder the development of motor skills, leading to reduced muscle force generation and decreased flexibility. Spastic cerebral palsy is the most prevalent type, affecting 77% of individuals with CP, and is caused by damage to the motor cortex and pyramidal tracts. The motor cortex is responsible for transmitting voluntary movement signals from the brain to the muscles. Characteristics of spastic cerebral palsy include stiff muscles (hypertonia), which can cause jerky and repetitive limb movements (spasticity). Additionally, individuals with CP often have difficulties in processing somatosensory and proprioceptive information. Proprioceptive training refers to interventions aimed at enhancing proprioceptive function to ultimately improve motor performance, a concept that has been explored in studies focused on sports injuries. In this study, we will utilize two proprioceptive exercises-rhythmic stabilization and ball balancing-to promote functional improvement in the upper extremities of children with spastic CP.

DETAILED DESCRIPTION:
There will be two groups: Group A will consist of 16 patients undergoing rhythmic stabilization, while Group B will also have 16 patients participating in ball balancing activities. Data will be collected both before and after the intervention to determine the most effective approach. Data analysis will be conducted using SPSS version 23.00.

This study will be a randomized clinical trial, with data collected from the University of Lahore Teaching Hospital (ULTH) and the Pakistan Society for the Rehabilitation of the Disabled (PSRD) in Lahore. A total of 32 patients will participate, equally divided into two groups through random allocation. The inclusion criteria will consist of children aged 5-12 with spastic CP, encompassing both genders. Patients with any neurological conditions, other orthopedic issues, a history of spine surgery, severe systemic disorders, psychiatric disorders, or neuromuscular disorders will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Spastic diplegic CP children age 6 to 12 years,
* Each gender included
* Grade 1 of spasticity according to modified Ashworth scale (21)
* With normal I.Q. greater than 70 (assessed by psychologist),
* Can follow commands(

Exclusion Criteria:

* Children with any other neurological impairment
* Children with audio visual impairment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
QUEST ( Quality of Upper Extremity Skills Test) | 6 weeks
  The Quality of Upper Extremity Skills Test (QUEST) is a reliable and valid tool that assesses hand function and movement patterns in children with cerebral palsy. It can be used with children aged 6 to 12 years (23). The test is conducted in a play environment and consists of 34 activity items. The test assesses four domains: Dissociated movements, Grasp, Protective extension. Reliability is 0.96 and validity is 0.84.
SHUEE Scale | 6 weeks
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function in children with hemiplegic cerebral palsy. This tool includes spontaneous functional analysis and Effects of Rhythmic Stabilization versus Ball Balancing on Spastic CP 3dynamic positional analysis and assesses the ability to perform grasp and release. The validity is 0.47 and reliability is 0.99

CONTACTS AND LOCATIONS:
Overall Officials: Masifah Kashif, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel DR, Neelakantan M, Pandher K, Merrick J. Cerebral palsy in children: a clinical overview. Transl Pediatr. 2020 Feb;9(Suppl 1):S125-S135. doi: 10.21037/tp.2020.01.01. PMID 32206590